CLINICAL TRIAL: NCT02713555
Title: Effects of Hepatic Insulin Resistance on Type 2 Diabetes Mellitus in Morbidly Obese Subjects Following Roux-en-Y Gastric Bypass Surgery or Gastric Sleeve Surgery
Brief Title: Effect of Roux-en-Y Gastric Bypass or Gastric Sleeve Surgery on Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYGBGS2016
Record Dates: First submitted 2016-03-04; First posted 2016-03-18 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Gastric Bypass; Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Roux-en-Y Gastric Bypass group (Experimental): Morbidly obese patients with type 2 diabetes mellitus will be examined before and after the Roux-en-Y Gastric Bypass procedure
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Gastric sleeve group (Experimental): Morbidly obese patient with type 2 diabetes Mellitus will be examined before and after the Gastric Sleeve procedure
  Interventions: Procedure: Gastric Sleeve
- Method /control group (No Intervention): Healthy normal weight participants matched by age and gender to the intervention study will be examined with the same methods as the intervention groups and serve as participants in a method study and as a metabolic normal reference group.

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — Roux-en-Y Gastric Bypass surgery entails the formation of a small gastric pouch and the division of the small intestine 60 cm from the duodenum. Formation of a gastrojejunal anastomosis with the distal segment and the formation of a jejuno-jejunal anastomosis 150 cm from the gastrojejunal anastomosis with the biliary segment.
  Other Names: Gastric Bypass
  Arms: Roux-en-Y Gastric Bypass group
Procedure: Gastric Sleeve — Gastric Sleeve entails a vertical division of the stomach with a stapler.
  Other Names: Gastrectomy
  Arms: Gastric sleeve group

SUMMARY:
Roux-en-Y Gastric Bypass surgery (RYGB) ameliorates type 2 diabetes within days after surgery. Studies indicate that the gastric sleeve procedure has comparable effect on type 2 diabetes, but to what extent and how is not fully elucidated. This study investigates the effect of the surgeries on incretin levels, glucose effectiveness and hepatic insulin sensitivity.

DETAILED DESCRIPTION:
Introduction This study comprises of a series of studies in morbidly obese subjects with type 2 diabetes before and after Roux-en-Y Gastric Bypass surgery (RYGB) and the gastric sleeve procedure, investigating the effect of these surgeries on incretin levels and hepatic insulin sensitivity. The method study (study 2) seeks to validate a better and physiological method to investigate insulin sensitivity in morbidly obese patients.

RYGB is considered the most effective treatment for obesity. The procedure improves glycemic control, and patients with type 2 diabetes may experience reductions in antidiabetic medication within days after surgery.

The improvement in glucose tolerance is associated with enhanced insulin action in muscle and adipose tissues. Recent reports indicate that hepatic insulin resistance also is improved, but the contribution of increased hepatic insulin action on glucose tolerance is controversial and remains to be thoroughly investigated. Studies indicate that RYGB reduces basal glucose production, and at 1 week following surgery hepatic insulin resistance is improved and insulin clearance increased. In contrast, insulin sensitivity in extra-hepatic tissues is not increased until 3 months after surgery. These observations imply that the liver plays an important role for early improvements in carbohydrate metabolism after RYBG, while increased insulin sensitivity in extra-hepatic tissues (muscle and adipose tissues) is delayed and more closely related to weight loss.

Effects of hepatic insulin sensitivity on glucose tolerance in obese subjects has in previous studies been addressed. However, dose response curves that determines time-dependent changes in hepatic insulin action are important for understanding the pathophysiology of glucose intolerance in obese subjects after RYGB, have not yet been conducted.

The development of a valid easy procedure that estimates insulin sensitivity at the same time the effect of the incretin hormones can be studied is of great value in especially RYGB operated patients where the secretion of hormones has been altered by the procedure. Understanding the impact of incretin hormones and hepatic insulin resistance on glucose intolerance may have implications for the medical treatment of obese patients, and may potentially predict which subset of patients are likely to experience the greatest benefits of RYGB or gastric sleeve surgery.

Moreover, a recent report indicates that the gastric sleeve procedure, where the stomach is reduced in size, elicits the same incretin response as RYGB, although no gastro-entero or entero-entero anastomosis are formed. Also the procedure is reported to have a profound effect on glucose intolerance. The mechanisms behind this have not yet been clarified.

Elucidation of these mechanisms will provide knowledge about body weight regulation and the pathophysiology of type 2 diabetes, and could help to identify new drug targets, improved study methods and surgical techniques.

The aims of the proposed PhD experiments are as follows:

Study 1.

1. To determine the contribution of hepatic insulin resistance to glucose intolerance in morbidly obese subjects
2. To examine to what extent increased hepatic insulin sensitivity contributes to normalization of glucose intolerance after RYGB and the gastric sleeve procedure.
3. Determine metabolic markers of defects in carbohydrate metabolism that may help to identify which patients are likely to benefit from RYGB or gastric sleeve. Indices will be determined based on a modified minimal model analysis of oral glucose tolerance test (OGTT) data.

Study 2.

1. To determine whether the minimal model behind the dynamic estimates of the OGTT can be further developed by simple addition of the two 2 tracer technique, when compared with data from the IVGTT and two step euglycaemic hyperinsulinaemic glucose clamp.

Experimental design

Study 1: The first of the proposed series of experiments attempts to determine how RYGB and the gastric sleeve procedure improves hepatic insulin resistance and if so how this affects glucose intolerance.

The study protocol is comprised of

1. An insulin-modified oral glucose tolerance test (OGTT) or a standard oral glucose tolerance test with double stable isotope tracer.
2. An insulin-modified intravenous glucose tolerance test (IVGTT) with radioactive tracer.
3. A hyperinsulinaemic euglycaemic glucose clamp with radioactive tracer.

The OGTT, IVGTT and the euglycaemic hyperinsulinaemic glucose clamp will be performed, prior to RYGB/gastric sleeve (usual care) and at 1, and 12 months following surgery (after intervention).

Liver biopsy will be performed at surgery, to assess liver steatosis and the effect of the obesity on liver insulin resistance and clearance. The effect over time of RYGB and gastric sleeve surgery will be assessed through secondary markers of liver function.

Study 2: The method study will be conducted in order to compare the indices from the two tracer OGTT to the euglycaemic hyperinsulinaemic glucose clamp and the insulin-modified intravenous glucose tolerance test to assess the estimates of insulin sensitivity and insulin clearance. The subjects will also serve as a normal metabolic reference group for study 1.

The study protocol is comprised of

1. An insulin-modified oral glucose tolerance test (OGTT) with double stable isotope tracer.
2. An insulin-modified intravenous glucose tolerance test (IVGTT) with radioactive tracer.
3. A hyperinsulinaemic euglycaemic glucose clamp with radioactive tracer.

For study 1 and 2

Indirect calorimetry will be assessed to determine changes in non-oxidative glucose disposal.

Dual energy X-ray absorptiometry (DEXA) scans will be performed to assess changes in fat and fat-free mass.

Sample size calculation

A sample size calculation has been performed to determine the number of study subjects required to obtain a statistical difference between groups. The calculation was performed based on the mean and standard deviation of the area above baseline calculation of glucose concentrations obtained during an OGTT in healthy subjects i.e. 290±217 mmol/L x min. The calculation was performed based on the following assumptions:

1. A difference in glucose tolerance in healthy controls and obese study subjects during the OGTT of 90% (unpaired analysis) and an improvement in glucose tolerance at 12 months after surgery in obese subjects of 50% (paired analysis)
2. Power of the analysis: 80%
3. Level of significance: 5% Based on these assumptions the sample size calculations require that 9 healthy subjects and 9 obese subjects undergoing RYGB or gastric sleeve need to successfully complete the full study program. To correct for an anticipated dropout rate during the studies a total of 12 obese for each surgical group and 12 healthy subjects will be recruited for the studies.

Materials and Calculations

A biobank will be opened at V laboratory Aarhus University hospital in an appropriate freezer. The material will be analyzed in small batches in order to avoid inter assay differences. The liver biopsy will be examined for histology the same day. After the project has come to an end any leftover material (blood or tissue) will be placed in a biobank for further research, should this prove valid and the research subject accept. Urine samples will be analyzed immediately and not preserved.

The oral glucose and C-peptide minimal model analysis of the OGTT data will yield indices for insulin sensitivity, beta-cell function (dynamic and static component), glucose effectiveness and hepatic insulin extraction. The disposition index i.e. the product of insulin sensitivity and beta cell function will be calculated.

Tracer determined rates of glucose production and uptake will be calculated using the equations for non-steady state. The volume of distribution of glucose will be assumed to be 200 ml/kg and a pool correction factor of 0.65 will be used in the calculations. Glucose specific activity will be calculated as the ratio between the tracer contraction and the prevailing plasma glucose concentration. The Hot Ginf technique will be used to maintain constant specific activities throughout the studies.

Side effect and risks

The patients and the metabolic controls subject will be exposed to radiation from the examinations.

The study subjects will be exposed to some radiation which will enhances their risk for a non-curable cancer from 25% to 25,005%.

Total amount of blood drawn 3-6 months prior to surgery is approximately 392 ml. Blood loss during surgery amounts to no more than 10-20 ml in general. Should complications such as infection or bleeding arise following surgery the patient will be excluded from the study. In the case of a minor perioperative bleeding the patient will be treated and observed according to surgical principles and the following study days 1 month later postponed if necessary.

Between 1 and 3 months after surgery 356 ml blood will be drawn. The patient will again be examined 12 months after surgery and 383 ml blood is drawn including blood samples for the endocrinology follow up-visit. All patients are substituted with iron and B12 vitamin from inclusion in the study and will prior to studies be examined with a spot hemoglobin (HB). Should the HB < 6,5 mmol/ l the study will be postponed for 3-5 weeks.

The liver biopsy during surgery leads to a minimal enhanced risk for bleeding and gall leak perioperative, but does not enhance the risk of the surgery in general. After the operation patients with type 2 diabetes are observed in the anesthesia postoperative ward and when ready (blood pressure, heart rate and pain under control) transferred to the surgical department for the first 24 hours and will here also be observed for changes in vital parameters.

Compensation will be provided in accordance with the guidelines from the local ethics committee.

Statistical analysis

When appropriate a paired Student's t test will be used to test for statistical difference. A non-parametric two sample analysis will be used for data not fulfilling the criteria for normal distribution. P < 0.05 will be considered statistically significant. ANOVA analysis aiming to detect difference in metabolic response between groups will be performed when appropriate.

Multivariate analysis will be performed to determine which indices are likely to be associated with the most favorable outcome. The analysis will be performed to assess which subset of obese subjects are most likely to benefit from the surgical procedure

Perspective

The above study plan will shed new light on the livers impact on diabetes, obesity and the significant effect of RYGB and gastric sleeve surgery on blood sugar control. The gastric sleeve surgery entails less risk for complications during and after surgery, should the procedure show comparable results with RYGB it can potentially benefit more patients planned for bariatric surgery. We also aim to validate an easy conductible and physiological method for obtaining reliable estimates of glucose kinetics. This can potentially lead to more specific diagnosis of for instance pancreatic islet cell function or hepatic insulin resistance, and thereby improve medical treatment of type 2 diabetes. The study also aims to identify biomarkers that can help to predict, which patients will benefit the most RYGB and gastric sleeve surgery.

All result, positive, negative or inconclusive will be published. We expect, at minimum to produce 4 articles, which will be accepted at international recognized magazines and 1 PhD thesis

Ethical aspects

The study is comprised of validated methods. Overall society, patients and future patient will benefit from the new insights into liver physiology in the state of obesity and diabetes before and after bariatric surgery. Future patients will also benefit from the new insights into the effects of the gastric sleeve surgery that entails less risk for complications. This can lead to improved treatments and more carefully selection of patient elective for surgery. The overall benefits for patients, future patients and society outweigh the risk and side effects the subjects endure.

The Danish data agency has approved the study and the regional ethics committee is processing the application.

Study completion

The proposed studies will be performed in collaboration between Hospital Unit Midt, Department of General Surgery where RYGB and gastric sleeve is performed. The glucose clamp studies will be performed at The Medical Research Lab, Departments of Medicine M and V, Aarhus University Hospital. All studies will be performed or supervised by PhD student Katrine Brodersen or Doctor of Medical Science Michael Festersen Nielsen.

Funding

All costs not covered by ongoing external funding will be covered by Hospital Unit Midt. Neither the PhD student nor the supervisor have any relations with the private foundations and nothing to declare.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 kg/m2
* Diabetes Mellitus, type 2

Exclusion Criteria:

* Diabetes Mellitus, type 1
* Chronic obstructive lung disease
* Heart failure or other cardiac disease
* Chronic inflammatory diseases
* Hepatitis or HIV
* Anemia
* Abnormal kidney or liver function
* Metabolic disease
* Prescription of prednisolone as pill or injection in the study period or 3 months prior to study start
* Alcoholism or abuse of other substances
* Pregnancy or planning to get pregnant within the study period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline diabetes status at 1 month after surgery | Baseline and 1 month
  fasting plasma glucose < 7.0 mmol/l
Change from baseline diabetes status at 12 months after surgery | Baseline and 12 months
  fasting plasma glucose < 7.0 mmol/l

SECONDARY OUTCOMES:
Weight loss from baseline | Baseline to 12 months
  Excess Body weight loss (%)
Weight loss from baseline | Baseline to 1 month
  Excess Body weight loss (%)
Estimates of changes in Insulin secretion from baseline | Baseline to 1 month
  Obtained through an oral glucose tolerance test and the minimal model
Estimates of changes in Insulin secretion from baseline | Baseline to 12 months
  Obtained through an oral glucose tolerance test and the minimal model
Estimates of changes in glucose effectiveness from baseline | Baseline to 1 month
  Obtained through an OGTT/IVGTT and the minimal model
Estimates of changes in glucose effectiveness from baseline | Baseline to 12 months
  Obtained through an OGTT/IVGTT and the minimal model
Estimates of changes in insulin clearance from baseline | Baseline to 1 month
  Obtained through an IVGTT and the minimal model
Estimates of changes in insulin clearance from baseline | Baseline to 12 months
  Obtained through an IVGTT and the minimal model
Estimates of changes in endogen glucose production from baseline | Baseline to 1 month
  Obtained through a two-step hyperinsulinaemic euglycaemic clamp
Estimates of changes in endogen glucose production from baseline | Baseline to 12 months
  Obtained through a two-step hyperinsulinaemic euglycaemic clamp
Assessment of Liver steatosis | 4 months
  Perioperative liver biopsy
Estimates of changes in Non-oxidative glucose-disposal from baseline | Baseline to 1 month
  Assessed through indirect calorimetry
Estimates of changes in Non-oxidative glucose-disposal from baseline | Baseline to 12 months
  Assessed through indirect calorimetry
Assessment og changes in fat and fat free mass from baseline | Baseline to 1 month
  Assessed through DEXA scan
Assessment og changes in fat and fat free mass from baseline | Baseline to 12 months
  Assessed through DEXA scan
Estimates of changes in insulin secretion from baseline | Baseline to 1 month
  Disposition index obtained through OGTT and the minimal model
Estimates of changes in insulin secretion from baseline | Baseline to 12 months
  Disposition index obtained through OGTT and the minimal model
Estimates of changes in insulin sensitivity from baseline | Baseline to 1 month
  Disposition index obtained through OGTT and the minimal model
Estimates of changes in insulin sensitivity from baseline | Baseline to 12 months
  Disposition index obtained through OGTT and the minimal model
Assessment of changes in glucagon-like peptide-1 from baseline | Baseline to 1 month
  Blood samples: glucagon-like peptide obtained during an OGTT
Assessment of changes in glucagon-like peptide-1 from baseline | Baseline to 12 months
  Blood samples: glucagon-like peptide obtained during an OGTT
Assessment of changes in gastric inhibitor polypeptide from baseline | Baseline to 1 month
  Blood samples: gastric inhibitor polypeptide obtained during an OGTT
Assessment of changes in gastric inhibitor polypeptide from baseline | Baseline to 12 months
  Blood samples: gastric inhibitor polypeptide obtained during an OGTT
Assessment of changes in liver function from baseline | Baseline to 1 month
  Blood samples: Alanine Amino Transferase
Assessment of changes in liver function from baseline | Baseline to 12 months
  Blood samples: Alanine Amino Transferase
Assessment of changes in Ghrelin from baseline | Baseline to 1 month
  Blood samples: Ghrelin obtained during an OGTT
Assessment of changes in Ghrelin from baseline | Baseline to 12 months
  Blood samples: Ghrelin obtained during an OGTT
Assessment of changes in Leptin from baseline | Baseline to 1 month
  Blood samples: Leptin
Assessment of changes in Leptin from baseline | Baseline to 12 months
  Blood samples: Leptin
Assessment of the role of FGF21 in type 2 diabetes and obesity from baseline | Baseline to 1 month
  Blood sample: Fibroblast growth factor 21 (FGF21) obtained during an OGTT
Assessment of the role of FGF21 in type 2 diabetes and obesity from baseline | Baseline to 12 months
  Blood sample: Fibroblast growth factor 21 (FGF21) obtained during an OGTT
Assessment of changes in Glucagon levels from baseline | Baseline to 1 month
  Blood samples: glucagon obtained during an OGTT
Assessment of changes in Glucagon levels from baseline | Baseline to 12 months
  Blood samples: glucagon obtained during an OGTT

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Brodersen, PhD student, Principal Investigator — University of Aarhus, Hospital Unit Midt; Michael F. Nielsen, DMSc., Study Director — University of Aarhus, Hospital Unit Midt
Locations (1):
- Hospital Unit Midt, Viborg, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized transfer of data after study completion to the Danish Archive.

REFERENCES:
- [Background] Madsbad S, Dirksen C, Holst JJ. Mechanisms of changes in glucose metabolism and bodyweight after bariatric surgery. Lancet Diabetes Endocrinol. 2014 Feb;2(2):152-64. doi: 10.1016/S2213-8587(13)70218-3. Epub 2014 Feb 3. PMID 24622719
- [Background] Coppini LZ, Bertevello PL, Gama-Rodrigues J, Waitzberg DL. Changes in insulin sensitivity in morbidly obese patients with or without metabolic syndrome after gastric bypass. Obes Surg. 2006 Nov;16(11):1520-5. doi: 10.1381/096089206778870030. PMID 17132419
- [Background] Wellford AL, Snoey ER. Emergency medicine applications of echocardiography. Emerg Med Clin North Am. 1995 Nov;13(4):831-54. PMID 7588192
- [Background] Wickremesekera K, Miller G, Naotunne TD, Knowles G, Stubbs RS. Loss of insulin resistance after Roux-en-Y gastric bypass surgery: a time course study. Obes Surg. 2005 Apr;15(4):474-81. doi: 10.1381/0960892053723402. PMID 15946424
- [Background] Dirksen C, Jorgensen NB, Bojsen-Moller KN, Jacobsen SH, Hansen DL, Worm D, Holst JJ, Madsbad S. Mechanisms of improved glycaemic control after Roux-en-Y gastric bypass. Diabetologia. 2012 Jul;55(7):1890-901. doi: 10.1007/s00125-012-2556-7. Epub 2012 Apr 27. PMID 22538359
- [Background] Bojsen-Moller KN, Dirksen C, Jorgensen NB, Jacobsen SH, Serup AK, Albers PH, Hansen DL, Worm D, Naver L, Kristiansen VB, Wojtaszewski JF, Kiens B, Holst JJ, Richter EA, Madsbad S. Early enhancements of hepatic and later of peripheral insulin sensitivity combined with increased postprandial insulin secretion contribute to improved glycemic control after Roux-en-Y gastric bypass. Diabetes. 2014 May;63(5):1725-37. doi: 10.2337/db13-1307. Epub 2013 Nov 15. PMID 24241533
- [Background] Romero F, Nicolau J, Flores L, Casamitjana R, Ibarzabal A, Lacy A, Vidal J. Comparable early changes in gastrointestinal hormones after sleeve gastrectomy and Roux-En-Y gastric bypass surgery for morbidly obese type 2 diabetic subjects. Surg Endosc. 2012 Aug;26(8):2231-9. doi: 10.1007/s00464-012-2166-y. PMID 22302537
- [Background] Nielsen MF, Caumo A, Aagaard NK, Chandramouli V, Schumann WC, Landau BR, Schmitz O, Vilstrup H. Contribution of defects in glucose uptake to carbohydrate intolerance in liver cirrhosis: assessment during physiological glucose and insulin concentrations. Am J Physiol Gastrointest Liver Physiol. 2005 Jun;288(6):G1135-43. doi: 10.1152/ajpgi.00278.2004. Epub 2005 Jan 6. PMID 15637182
- [Background] Dalla Man C, Caumo A, Basu R, Rizza R, Toffolo G, Cobelli C. Minimal model estimation of glucose absorption and insulin sensitivity from oral test: validation with a tracer method. Am J Physiol Endocrinol Metab. 2004 Oct;287(4):E637-43. doi: 10.1152/ajpendo.00319.2003. Epub 2004 May 11. PMID 15138152
- [Background] Dalla Man C, Caumo A, Basu R, Rizza R, Toffolo G, Cobelli C. Measurement of selective effect of insulin on glucose disposal from labeled glucose oral test minimal model. Am J Physiol Endocrinol Metab. 2005 Nov;289(5):E909-14. doi: 10.1152/ajpendo.00299.2004. Epub 2005 Jun 21. PMID 15972269
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] STEELE R, WALL JS, DE BODO RC, ALTSZULER N. Measurement of size and turnover rate of body glucose pool by the isotope dilution method. Am J Physiol. 1956 Sep;187(1):15-24. doi: 10.1152/ajplegacy.1956.187.1.15. No abstract available. PMID 13362583
- [Derived] Visentin R, Brodersen K, Richelsen B, Moller N, Dalla Man C, Pedersen AK, Abrahamsen J, Holst JJ, Nielsen MF. Increased Insulin Secretion and Glucose Effectiveness in Obese Patients with Type 2 Diabetes following Bariatric Surgery. J Diabetes Res. 2023 Nov 14;2023:7127426. doi: 10.1155/2023/7127426. eCollection 2023. PMID 38020201
- [Derived] Brodersen K, Nielsen MF, Richelsen B, Lauritzen ES, Pahle E, Abrahamsen J, Hartmann B, Holst JJ, Moller N. Comparable Effects of Sleeve Gastrectomy and Roux-en-Y Gastric Bypass on Basal Fuel Metabolism and Insulin Sensitivity in Individuals with Obesity and Type 2 Diabetes. J Diabetes Res. 2022 Dec 21;2022:5476454. doi: 10.1155/2022/5476454. eCollection 2022. PMID 36589629